CLINICAL TRIAL: NCT03171558
Title: Gastric Pull up Versus Free Flaps Reconstruction (Anterolateral Thigh and Radial Forearm Free Flap) for Laryngo-pharyngeal Defects: A Prospective Randomized Trial
Brief Title: Gastric Pull up Versus Free Flap Reconstruction for Laryngo-pharyngeal Defects
Acronym: GPU vs ALT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Eitan Prisman, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H14-00004
Record Dates: First submitted 2017-02-22; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Neoplasms; Pharyngectomy; Reconstructive Surgical Procedures
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric Pull Up (Experimental): Patients randomized to undergo gastric pull up surgical reconstruction of pharyngoesophageal defect.
  Interventions: Procedure: Gastric Pull Up
- Free Flap (Active Comparator): Patients randomized to undergo free flap (anterolateral thigh or radial forearm) surgical reconstruction of pharyngoesophageal defect.
  Interventions: Procedure: Free Flap Surgery

INTERVENTIONS:
Procedure: Gastric Pull Up — Using gastric tissue to reconstruct the esophagus and pharynx after pharyngo-esophagectomy.
  Arms: Gastric Pull Up
Procedure: Free Flap Surgery — Using radial forearm free flap or anterolateral thigh free flap to reconstruct the cervical esophagus and pharynx after pharyngectomy and cervical esophagectomy.
  Other Names: Anterolateral thigh free flap and radial forearm free flap
  Arms: Free Flap

SUMMARY:
This study will compare the gastric pull up (GPU) with the free flap [(specifically, anterolateral thigh (ALT) and radial forearm free flap (RFFF)] techniques used in the reconstruction of alimentary tracts in patients who require laryngectomy and circumferential pharyngectomy for carcinoma resection. These two interventions will be compared by block randomizing 20 patients based on history of failed chemoradiation to undergo either ALT or RFFF. The primary outcome will be the type and number of postoperative complications. The secondary outcomes will include swallowing function, speech, and quality of life measures along with cancer specific endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent, attend follow-up visits and complete questionnaires
* Have an Eastern Cooperation Oncology Group (ECOG) performance status of 0-2
* Patients with carcinoma of thyroid, larynx, hypopharynx, or cervical esophagus requiring surgery as a primary treatment modality or after chemoradiation treatment failure
* Laryngectomy and circumferential pharyngectomy as recommended by the head and neck tumor board

Exclusion Criteria:

* Serious medical co morbidities or other contraindications to surgery
* Metastatic disease
* Pregnant or lactating women
* Patients whose clinical circumstances are such that one surgical intervention would be recommended over the other: The cancer extends into the the thorax as seen on pre-operative CT scan. In these patients, the GPU reconstruction is preferred.
* Patients who have liver cirrhosis or multiple previous surgeries on the stomach would not be candidates for the GPU and thus will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Type and number of postoperative complications | Within 90 days of surgery occurring on the same or separate admission.
  Complications will be divided by: (1) in-hospital mortality (2) reconstruction related complications (anastomotic leak, fistula formation, flap necrosis, flap stenosis or stricture, requirement for surgical revision), and (3) addition in-hospital complications ( bleeding, pulmonary, cardiac, infectious, abdominal, wound concern)

SECONDARY OUTCOMES:
Surgical Time | Initial Surgery
  Time from first incision to the end of surgical closure as documented on the nursing record.
Operative blood loss | Initial surgery
  Total volume of blood lost and accounted for in suction canisters as documented in nursing charts. (this excludes blood not accounted for in the suction containers)
Operative Parameters | During initial surgery and within the first 72 hours.
  Requirement for transfusion, measured in units of blood.
Flap Donor Site Morbidity (RFFF) ) | Measure documented at 1, 3, 6 and 12 months post-surgery, thereafter yearly for 5 years. (8 visits total)
  Donor site associated quality of life (Toronto Extremity Salvage Score - Upper Extremity)
Flap Donor Site Morbidity (ALT) | Measure documented at 1, 3, 6 and 12 months post-surgery, thereafter yearly for 5 years. (8 visits total)
  Donor site associated quality of life (Toronto Extremity Salvage Score - Lower Extremity)
Time to return to swallowing | If occurs in hospital will be documented by the treating team. Otherwise will be documented based on patient or speech language pathology reporting at 1, 3, 6 and 12 months post-surgery, thereafter yearly for 5 years. (9 visits total)
  Time from surgery to swallowing liquids.
Time to return of FULL oral diet | Measure documented at 1, 3, 6 and 12 months post-surgery, thereafter yearly for 5 years. (9 visits total)
  Time from surgery to return of diet that is sufficient for patient to maintain nutrition without requiring G-tube or NG feeding. Patient or Speech Language Pathology reported.
Requirement for feeding tube at 1 year after surgery. | Documented at 1 year follow up visit.
  Whether patients are still feeding tube dependent for nutrition at 1 year follow up.
Voice Function | Measure documented at time of surgical booking and at 1, 3, 6 and 12 months post-surgery, thereafter yearly for 5 years. (9 visits total)
  Measured by Voice Handicap Index -10
Dysphagia | Measure documented at time of surgical booking and at 1, 3, 6 and 12 months post-surgery, thereafter yearly for 5 years. (9 visits total)
  M.D. Anderson Dysphagia Inventory for assessment of dysphagia
Dumping Symptoms | Measure documented at time of surgical booking and at 1, 3, 6 and 12 months post-surgery, thereafter yearly for 5 years. (9 visits total)
  Assessed with the dumping symptom rating scale
Quality of Life | Measure documented at 1, 3, 6 and 12 months post-surgery, thereafter yearly for 5 years. (8 visits total)
  Measure with combined scores of two questionnaires: European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ) - C30 and EORTC QLQ - H&N35
Margin status of the resected specimen as reported by pathology | At the time of surgery
  Will be classified as positive and negative based on what is reported at Vancouver General Hospital Pathology reports generated at the time of surgery. A measure of clearance in millimeters will also be provided.
Time to progression | Patients will be monitored for 5 years post-operatively
  time from the date of the surgery until local, regional, or metastatic disease is detected
Disease Free Survival | Patients will be monitored for 5 years post-operatively
  Time from the date of the surgery until a patient experiences a recurrence, a new primary cancer or death
Progression-free survival | Patients will be monitored for 5 years post-operatively
  Time from the date of the surgery until a patient shows sign of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Prisman Eitan, MD, FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.